CLINICAL TRIAL: NCT01282476
Title: Panobinostat in Combination With Rituximab For Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: Panobinostat With Rituximab for Relapsed/Refractory Diffuse Large B Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-441
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-04

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL (Diffuse Large B Cell Lymphoma); Panobinostat; LBH589 (Panobinostat); LBH-589 (Panobinostat); HDAC inhibitor (Histone deacetylase inhibitor); DAC inhibitor (deacetylase inhibitor); deacetylase inhibitor; lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating; Lymphoma | interventions — Panobinostat; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panobinostat/Rituximab (Experimental): single-arm, open-label; Panobinostat with Rituximab: Panobinostat 40 mg orally 3 x weekly Rituximab 375 mg/m^2 IV days 1,8,15,and 22 of cycle 1, and then on day 1 of subsequent cycles.
  Interventions: Drug: Panobinostat with Rituximab

INTERVENTIONS:
Drug: Panobinostat with Rituximab — Panobinostat 40 mg orally 3 x weekly Rituximab 375 mg/m^2 IV days 1,8,15,and 22 of cycle 1, and then on day 1 of subsequent cycles.
  Other Names: LBH589; LBH-569; Rituxan

SUMMARY:
Panobinostat is a drug that may slow down the growth of cancer cells or kill cancer cells by blocking certain enzymes. Panobinostat has shown effects against cancer in laboratory studies. However, it is not known if it will show the same activity in humans. Panobinostat has been given to participants with various types of cancers, including DLBCL, in previous research studies. In this study panobinostat will be given with the the antibody rituximab, which is FDA approved to be given with chemotherapy in DLBCL.

DETAILED DESCRIPTION:
Study treatment will be given in 4 week periods called cycles. Panobinostat will be taken orally on Monday, Wednesday, and Friday of each week. Rituximab will be given as an intravenous infusion weekly during Cycle 1 and then once per month on day 1 of subsequent cycles. Subjects can receive up to 6 cycles of treatment. Blood draws and 2 EKGs (electrocardiograms) will be done weekly in Cycle 1 and then once in each cycle. PET/CT (Positron Emission Tomography/Computed Tomography) scans will be done every 2 months.

If disease has not progressed after 6 cycles on combination of panobinostat and rituximab, subjects may continue on panobinostat alone for up to 6 additional months.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory DLBCL
* More than 1 line of prior chemotherapy

Exclusion Criteria:

* Currently receiving anticancer therapy or investigational agents
* Major surgery within last 4 weeks
* Known leptomeningeal or brain metastases
* Known HIV infection
* Uncontrolled fungal, bacterial, viral or other infection
* History of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least 3 years
* Hepatitis B or C positive
* GI disease
* Pregnant or breastfeeding
* Prior treatment with an HDAC inhibitor including valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panobinostat/Rituximab
Started | 18
Completed | 7
Not Completed | 11
Not completed — Death | 11

BASELINE CHARACTERISTICS:
Arm/Group | Panobinostat/Rituximab
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 68 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17
  Other | 1
Region of Enrollment [Number; unit: participants] — 8 from DFCI, 10 from MGH
  participants
    United States | 18
Histology [Count of Participants; unit: Participants]
  Centroblastic DLBCL(Diffuse large B cell lymphoma) | 1
  DLBCL follicular cell derivation w/high grade BCL | 1
  DLBCL not otherwise specified | 14
  DLBCL of follicular center derivation | 1
  Gray zone lymphoma | 1
EKG (electrocardiogram) [Count of Participants; unit: Participants]
  Abnormal | 3
  Normal | 15
elevated LDH (Lactate dehydrogenase) [Count of Participants; unit: Participants]
  Yes | 9
  No | 3
  Missing | 6
ECOG PS (Eastern Cooperative Oncology Group Performance Status) [Count of Participants; unit: Participants]
  00-Fully Active | 7
  01-Restricted | 8
  02-Ambulatory and Capable of Self Care | 3
Disease status [Count of Participants; unit: Participants]
  Refractory | 10
  Relapsed | 8
Number of extranodal sites [Count of Participants; unit: Participants]
  0 | 1
  1 | 3
  2 | 3
  3 | 9
  6 | 2
Number of target lesions [Count of Participants; unit: Participants]
  0-2 | 4
  3-5 | 6
  6+ | 8
Number of non-target lesions [Count of Participants; unit: Participants]
  0-2 | 12
  3-5 | 4
  6+ | 2
Time from last prior therapy [Median (Full Range); unit: days] | 117 [10 to 776]
Number of prior therapies [Count of Participants; unit: Participants]
  1-4 | 7
  5-8 | 9
  9+ | 2
Number of prior non-surgical therapies [Count of Participants; unit: Participants]
  0-2 | 6
  3-5 | 7
  6-8 | 5
Number of prior surgeries [Count of Participants; unit: Participants]
  0 | 12
  1 | 2
  2 | 2
  3 | 1
  4 | 1
Number of prior radiation treatments [Count of Participants; unit: Participants]
  0 | 12
  1 | 3
  2 | 2
  3 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is defined by the Revised International Workshop Response Criteria (2007) (see reference in protocol section).
  Overall response (OR) = Complete response (CR) + Partial response (PR)
Time Frame: 1 year
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Panobinostat/Rituximab
Number analyzed (Participants) | 18
percentage of participants | 11 [2 to 31]

2. Secondary Outcome: Progression-free Survival Rate
Description: Progression is defined by the Revised International Workshop Response Criteria (2007) (see reference in protocol section).
Time Frame: 6 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Panobinostat/Rituximab
Number analyzed (Participants) | 18
percentage of participants | 6 [0.7 to 21]

3. Secondary Outcome: Toxicities
Description: Evaluate safety of this combination in relapsed/refractory DLBCL patients Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat/Rituximab
Number analyzed (Participants) | 18
Participants
  Platelet count decreased: Grade 1 | 5
  Platelet count decreased: Grade 2 | 1
  Platelet count decreased: Grade 3 | 1
  Platelet count decreased: Grade 4 | 7
  Platelet count decreased: Did not have any | 4
  Fatigue: Grade 1 | 7
  Fatigue: Grade 2 | 1
  Fatigue: Grade 3 | 3
  Fatigue: Grade 4 | 0
  Fatigue: Did not have any | 7
  Anemia: Grade 1 | 3
  Anemia: Grade 2 | 3
  Anemia: Grade 3 | 4
  Anemia: Grade 4 | 0
  Anemia: Did not have any | 8
  Diarrhea: Grade 1 | 5
  Diarrhea: Grade 2 | 1
  Diarrhea: Grade 3 | 2
  Diarrhea: Grade 4 | 0
  Diarrhea: Did not have any | 10
  Nausea: Grade 1 | 5
  Nausea: Grade 2 | 0
  Nausea: Grade 3 | 0
  Nausea: Grade 4 | 0
  Nausea: Did not have any | 13
  Lymphocyte count decreased: Grade 1 | 0
  Lymphocyte count decreased: Grade 2 | 1
  Lymphocyte count decreased: Grade 3 | 3
  Lymphocyte count decreased: Grade 4 | 1
  Lymphocyte count decreased: Did not have any | 13
  Anorexia: Grade 1 | 4
  Anorexia: Grade 2 | 1
  Anorexia: Grade 3 | 0
  Anorexia: Grade 4 | 0
  Anorexia: Did not have any | 13
  Hypophosphatemia: Grade 1 | 2
  Hypophosphatemia: Grade 2 | 2
  Hypophosphatemia: Grade 3 | 0
  Hypophosphatemia: Grade 4 | 1
  Hypophosphatemia: Did not have any | 13
  Neutrophil count decreased: Grade 1 | 0
  Neutrophil count decreased: Grade 2 | 1
  Neutrophil count decreased: Grade 3 | 2
  Neutrophil count decreased: Grade 4 | 1
  Neutrophil count decreased: Did not have any | 14
  Hypoalbuminemia: Grade 1 | 4
  Hypoalbuminemia: Grade 2 | 0
  Hypoalbuminemia: Grade 3 | 0
  Hypoalbuminemia: Grade 4 | 0
  Hypoalbuminemia: Did not have any | 14
  Dyspnea: Grade 1 | 4
  Dyspnea: Grade 2 | 0
  Dyspnea: Grade 3 | 0
  Dyspnea: Grade 4 | 0
  Dyspnea: Did not have any | 14
  Constipation: Grade 1 | 3
  Constipation: Grade 2 | 0
  Constipation: Grade 3 | 0
  Constipation: Grade 4 | 0
  Constipation: Did not have any | 15
  Alkaline phosphatase increased: Grade 1 | 3
  Alkaline phosphatase increased: Grade 2 | 0
  Alkaline phosphatase increased: Grade 3 | 0
  Alkaline phosphatase increased: Grade 4 | 0
  Alkaline phosphatase increased: Did not have any | 15
  Creatinine increased: Grade 1 | 3
  Creatinine increased: Grade 2 | 0
  Creatinine increased: Grade 3 | 0
  Creatinine increased: Grade 4 | 0
  Creatinine increased: Did not have any | 15
  White blood cell decreased: Grade 1 | 0
  White blood cell decreased: Grade 2 | 0
  White blood cell decreased: Grade 3 | 2
  White blood cell decreased: Grade 4 | 1
  White blood cell decreased: Did not have any | 15
  Hypocalcemia: Grade 1 | 3
  Hypocalcemia: Grade 2 | 0
  Hypocalcemia: Grade 3 | 0
  Hypocalcemia: Grade 4 | 0
  Hypocalcemia: Did not have any | 15
  Hypokalemia: Grade 1 | 0
  Hypokalemia: Grade 2 | 0
  Hypokalemia: Grade 3 | 0
  Hypokalemia: Grade 4 | 2
  Hypokalemia: Did not have any | 16
  Hypomagnesemia: Grade 1 | 2
  Hypomagnesemia: Grade 2 | 0
  Hypomagnesemia: Grade 3 | 0
  Hypomagnesemia: Grade 4 | 0
  Hypomagnesemia: Did not have any | 16
  Dry mouth: Grade 1 | 1
  Dry mouth: Grade 2 | 0
  Dry mouth: Grade 3 | 0
  Dry mouth: Grade 4 | 0
  Dry mouth: Did not have any | 17
  Flatulence: Grade 1 | 1
  Flatulence: Grade 2 | 0
  Flatulence: Grade 3 | 0
  Flatulence: Grade 4 | 0
  Flatulence: Did not have any | 17
  Gatstroesophageal reflux disease: Grade 1 | 1
  Gatstroesophageal reflux disease: Grade 2 | 0
  Gatstroesophageal reflux disease: Grade 3 | 0
  Gatstroesophageal reflux disease: Grade 4 | 0
  Gatstroesophageal reflux disease: Did not have any | 17
  Mucositis oral: Grade 1 | 1
  Mucositis oral: Grade 2 | 0
  Mucositis oral: Grade 3 | 0
  Mucositis oral: Grade 4 | 0
  Mucositis oral: Did not have any | 17
  Vomiting: Grade 1 | 1
  Vomiting: Grade 2 | 0
  Vomiting: Grade 3 | 0
  Vomiting: Grade 4 | 0
  Vomiting: Did not have any | 17
  Edema face: Grade 1 | 1
  Edema face: Grade 2 | 0
  Edema face: Grade 3 | 0
  Edema face: Grade 4 | 0
  Edema face: Did not have any | 17
  Edema limbs: Grade 1 | 1
  Edema limbs: Grade 2 | 0
  Edema limbs: Grade 3 | 0
  Edema limbs: Grade 4 | 0
  Edema limbs: Did not have any | 17
  Fever: Grade 1 | 0
  Fever: Grade 2 | 1
  Fever: Grade 3 | 0
  Fever: Grade 4 | 0
  Fever: Did not have any | 17
  Hepatobiliary disorders - other: Grade 1 | 0
  Hepatobiliary disorders - other: Grade 2 | 0
  Hepatobiliary disorders - other: Grade 3 | 1
  Hepatobiliary disorders - other: Grade 4 | 0
  Hepatobiliary disorders - other: Did not have any | 17
  Aspartate aminotransferase increased: Grade 1 | 1
  Aspartate aminotransferase increased: Grade 2 | 0
  Aspartate aminotransferase increased: Grade 3 | 0
  Aspartate aminotransferase increased: Grade 4 | 0
  Aspartate aminotransferase increased: Did not have any | 17
  Blood bilirubin increased: Grade 1 | 1
  Blood bilirubin increased: Grade 2 | 0
  Blood bilirubin increased: Grade 3 | 0
  Blood bilirubin increased: Grade 4 | 0
  Blood bilirubin increased: Did not have any | 17
  Metabolism and nutrition disorders - other: Grade 1 | 0
  Metabolism and nutrition disorders - other: Grade 2 | 1
  Metabolism and nutrition disorders - other: Grade 3 | 0
  Metabolism and nutrition disorders - other: Grade 4 | 0
  Metabolism and nutrition disorders - other: Did not have any | 17
  Bone pain: Grade 1 | 1
  Bone pain: Grade 2 | 0
  Bone pain: Grade 3 | 0
  Bone pain: Grade 4 | 0
  Bone pain: Did not have any | 17
  Dysgeusia: Grade 1 | 1
  Dysgeusia: Grade 2 | 0
  Dysgeusia: Grade 3 | 0
  Dysgeusia: Grade 4 | 0
  Dysgeusia: Did not have any | 17
  Headache: Grade 1 | 1
  Headache: Grade 2 | 0
  Headache: Grade 3 | 0
  Headache: Grade 4 | 0
  Headache: Did not have any | 17
  Insomnia: Grade 1 | 1
  Insomnia: Grade 2 | 0
  Insomnia: Grade 3 | 0
  Insomnia: Grade 4 | 0
  Insomnia: Did not have any | 17
  Epistaxis: Grade 1 | 1
  Epistaxis: Grade 2 | 0
  Epistaxis: Grade 3 | 0
  Epistaxis: Grade 4 | 0
  Epistaxis: Did not have any | 17
  Skin and subcutaneous tissue disorders - other: Grade 1 | 0
  Skin and subcutaneous tissue disorders - other: Grade 2 | 0
  Skin and subcutaneous tissue disorders - other: Grade 3 | 1
  Skin and subcutaneous tissue disorders - other: Grade 4 | 0
  Skin and subcutaneous tissue disorders - other: Did not have any | 17

ADVERSE EVENTS:
Arm/Group | Panobinostat/Rituximab
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat/Rituximab (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Bilateral Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Death (General disorders) | 3 (3)
Death from disease progression (Blood and lymphatic system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Leukocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pain (back) (General disorders) | 1 (1)
Right lower extremity cellulitis (Infections and infestations) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panobinostat/Rituximab (N=18)
Platelet count decreased (Investigations) | 12 (30)
Fatigue (General disorders) | 13 (24)
Anemia (Blood and lymphatic system disorders) | 12 (29)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Lymphocyte count decrease (Investigations) | 7 (19)
Nausea (Gastrointestinal disorders) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Neutrophil count decrease (Investigations) | 4 (15)
Constipation (Gastrointestinal disorders) | 4 (6)
Edema limbs (General disorders) | 4 (4)
White blood cell decrease (Investigations) | 3 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Alkaline phosphatase increase (Investigations) | 3 (3)
Creatinine increased (Investigations) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Anxiety (Nervous system disorders) | 2 (2)
Blood bilirubin increase (Investigations) | 2 (2)
Pain (General disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuro (Nervous system disorders) | 2 (2)
Vascular disorders - Oth (Vascular disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Activated partial thromb (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransfera (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
General disorders (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hepatobiliary disorders (Hepatobiliary disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations - Other (Investigations) | 1 (1)
Metabolism and nutrition (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelitis (Nervous system disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropa (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No